CLINICAL TRIAL: NCT02251873
Title: An Open Label, Randomised, Parallel Group Study of the Drug-drug Pharmacokinetic Interaction of Steady State Tipranavir (SEDDS SEC) 500 mg and Ritonavir (Soft Gelatin Capsules) 100 mg or Tipranavir 750 mg and Ritonavir 200 mg, Both Bid for 13.5 Days With Single Dose Didanosine 400 mg (Delayed Release Capsule EC Beadlets) in Healthy Volunteers
Brief Title: Evaluation of the Pharmacokinetic Interaction of Steady State Tipranavir and Ritonavir or Tipranavir and Ritonavir With Single Dose Didanosine in Healthy Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 1182.42
Record Dates: First submitted 2014-09-25; First posted 2014-09-29 (Estimated); Last update posted 2014-09-29 (Estimated); Status verified 2014-09

CONDITIONS: Healthy
MeSH Terms: interventions — Ritonavir

ARMS (2):
- TPV + RTV (low dose)+ ddI (Experimental)
  Interventions: Drug: TPV + RTV (low dose); Drug: ddl
- TPV+ RTV (high dose)+ ddI (Experimental)
  Interventions: Drug: TPV + RTV (high dose); Drug: ddl

INTERVENTIONS:
Drug: TPV + RTV (low dose)
  Arms: TPV + RTV (low dose)+ ddI
Drug: TPV + RTV (high dose)
  Arms: TPV+ RTV (high dose)+ ddI
Drug: ddl

SUMMARY:
Study to characterise the effects of concurrent tipranavir (TPV) and ritonavir (RTV) administration on the single dose pharmacokinetics of didanosine (ddI), to characterise the effects of single-dose ddI on the pharmacokinetics of TPV and RTV and to assess the short-term safety of this combination

ELIGIBILITY:
Inclusion Criteria:

* Healthy male or female subjects as determined by results of screening
* Female subjects were not lactating and not of child bearing potential as defined by surgically sterile or post menopausal (no periods for at least 12 months and elevated follicle stimulating hormone (FSH) with low estradiol and no estrogen supplementation). Females were to use barrier contraception (e.g. condoms) for at least one month prior to administration of study medication, during the study and at least one month after release from the study. Women were to have negative pregnancy tests
* Signed written informed consent in accordance with Good Clinical Practice (GCP) and local legislation
* Age >=18 and <=60 years
* Body mass index (BMI) >=18.5 and <=29.9 kg/m2

Exclusion Criteria:

* Any finding of the medical examination (including blood pressure, pulse rate and ECG) deviating from normal and of clinical relevance
* History or current gastrointestinal, hepatic, renal, respiratory, cardiovascular, metabolic, immunologic, hormonal disorders, including a clinical history of viral hepatitis, or serological evidence of active Hepatitis B, Hepatitis C, or HIV infection
* History of orthostatic hypotension, fainting spells and blackouts
* Diseases of the central nervous system (such as epilepsy) or psychiatric disorders or neurological disorders
* Chronic or relevant acute infections
* History of allergy/hypersensitivity (including drug allergy) which was deemed relevant to the trial as judged by the investigator including study drugs
* Intake of drugs with a long half-life (> 24 hours) or enzyme altering drug within 1 month prior to administration of study drugs
* Use of any drugs that might have influenced the results of the trial within 10 days prior to administration or during the trial (in addition to specific medication prohibitions mentioned in exclusion criteria above)
* Use of grapefruit or grapefruit juice, alcohol, green tea, methylxanthine-containing products or tobacco within one week of study drug administration
* Participation in another trial with an investigational drug within 2 months prior to administration or during the trial
* Smoker (> 10 cigarettes or 3 cigars or 3 pipes/day) or inability to refrain from smoking on trial days
* Alcohol abuse (> 60 g/day)
* Drug abuse
* Blood or plasma donation within 1 month prior to administration or during the trial
* Excessive physical activities within 5 days prior to administration or during the trial
* Following specific laboratory findings: activated partial thromboplastin time (aPTT), prothrombin time international normalised ratio (INR), aspartate transaminase (AST), alanine transaminase (ALT), gamma-glutamyl-transferase (GGT), amylase, lipase, or triglyceride above the normal range
* Any other laboratory value outside the clinically accepted reference range and of clinical relevance
* History of any familial bleeding disorder
* Inability to swallow multiple large capsules
* Inability to comply with dietary regimen of study centre
* Inability to comply with investigator's instructions

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 50 (Actual)
Dates: Start 2001-09; Primary Completion 2002-03 (Actual)

PRIMARY OUTCOMES:
(AUC 0-12) Area under the plasma concentration time curve from 0-12 hours | up to 12 hours after dose administration
Cmax (Maximum measured concentration of the analyte in plasma) | up to 12 hours after dose administration
(C6h) drug concentration in plasma at 6 hours after drug administration | up to 6 hours after dose administration
(C12h) drug concentration in plasma at 12 hours after drug administration | up to 12 hours after dose administration
Cnh (plasma concentration n hours after drug administration) | up to 12 hours after dose administration

SECONDARY OUTCOMES:
Cmax,ss (maximum plasma concentration at steady state) | up to 12 hours after dose administration
MRT (mean residence time) | up to 12 hours after dose administration
Tmax (time to the maximum plasma concentration) | up to 12 hours after dose administration
CL/F (apparent oral clearance) | up to 12 hours after dose administration
Vz/F (apparent volume of distribution) | up to 12 hours after dose administration
t½ (Terminal half-life of the analyte in plasma) | up to 12 hours after dose administration
Number of subjects with adverse events | up to 40 days
Number of subjects with abnormal changes in laboratory parameters | up to 40 days